CLINICAL TRIAL: NCT06299943
Title: Blind Randomized Controlled Study of Biofeedback Training Based on Target Biomechanical Gait Parameters at Patients in the Early Recovery Period of Stroke Whith Hemiparesis
Brief Title: Biofeedback Gait Training by Target Biomechanical Parameters in the Early Recovery Period of Stroke
Acronym: TargetGait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BiofeedbackTargetGaitTraining
Record Dates: First submitted 2024-02-20; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Biofeedback; Gait, Hemiplegic; Gait Training; Hemiparesis
Keywords: stroke; hemiparesis; gait; rehabilitation; biofeedback
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Paresis

STUDY DESIGN:
Intervention Model Description: Parallel-group, single-blinded controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinicians involved in the measurements and researchers that worked with data results did not know which group each patient was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Target Biofeedbak gait training (Experimental): Patients in this group receive, in addition to conventional therapy, biofeedback gait training by selected biomechanical (Staince or single support phase, range of motion at joint or EMG amplitude) gait parameter. Training takes place 8-12 times over three weeks. The duration of each workout varies from 10 to 30 minutes.
  Interventions: Other: Biofeedback gait training by biomechanical target parameter
- Target Biofeedbak gait training-2 (Experimental): Patients in this group receive, in addition to conventional therapy, biofeedback gait training by selected biomechanical (Staince or single support phase, range of motion at joint or EMG amplitude) gait parameter. Training takes place 8-12 times over three weeks. The duration of each workout varies from 10 to 30 minutes.
  Interventions: Other: Biofeedback gait training by biomechanical target parameter

INTERVENTIONS:
Other: Biofeedback gait training by biomechanical target parameter — The patient walks using a treadmill at a comfortable speed until he gets tired. The patient is instructed that when performing a virtual task (in a virtual environment on the screen), his walking will be harmonized (without informing him on what parameter). If it fails to cope, then the zones of permissible changes (on the information columns) will expand, and the virtual task will signal its incomplete completion.

SUMMARY:
Single-blinded controlled clinical trial. Biofeedback training courses based on target biomechanical gait parameters are being studied. For targeted biofeedback training, various biomechanical parameters are used: parameters of the gait cycle, EMG or kinematics of joint movements. The number of sessions is 8-11 for each patient. Clinical gain analysis is carried out before and after a course of training. Changes in biomechanical parameters that occurred at the end of the training course are assessed in comparison with those before training, and both statuses (before and after training) are compared with similar gait parameters in a group of healthy adults.

DETAILED DESCRIPTION:
Walking function disorders are typical for patients after cerebral stroke. A cerebral stroke normally affects one hemisphere and causes a hemiplegic syndrome. The gait of hemiplegic patients has very specific features: reduced walking speed, increased double stance phase, and reduced amplitude of movement in the leg joints. Biofeedback technology (BFB) is currently considered effective and promising for training walking function, including in patients after cerebral stroke. The technology is based on capturing a physiological parameter and presenting it to the patient in a perceivable form, so that the subject can understand its changes and respond appropriately. BFB can be used independently or as part of rehabilitation therapy. Nevertheless, efficiency, as noted by most authors, remains the subject of discussion. This is due to the fact, that at the previous stage of development of these systems, there was no technical capability to use the specific biomechanical gait parameters as targets for training. Therefore, more general parameters-such as walking speed, step frequency, etc.-were and are still used. This circumstance is attributable to the very nature of the main biomechanical gait parameters, which require special means of recording. One of the significant technical difficulties in BFB implementation is the need for accurate and fast registration of the gait parameters in real-time to use them for biofeedback. At the same time, the use of portable sensors for BFB training goals can represent a certain solution to technical problems. In recent years, owing to its important advantages, wearable IMU technology (systems using inertial measurement units) has been widely applied for capturing biomechanical gait parameters. Investigators used a system that was originally developed with our participation for targeted training based on biofeedback according to the biomechanical parameters of gait. The use of inertial technology and artificial intelligence technology has made it possible to use biomechanical parameters of gait (time and general gait parameters, EMG and kinematics of leg's joints) for biofeedback in a very low-cost and practically convenient way. Biofeedback training courses based on target biomechanical gait parameters are being studied. For targeted biofeedback training, various biomechanical parameters are used: parameters of the gait cycle, EMG or kinematics of joint movements. The number of sessions is 8-11 for each patient. Clinical gait analysis is carried out before and after a course of training. Changes in biomechanical parameters that occurred at the end of the training course are assessed in comparison with those before training, and both statuses (before and after training) are compared with similar gait parameters in a group of healthy adults.

Stroke patients participated in the study in Federal Center of Cerebrovascular Pathology and Stroke FMBA in Moscow, Russia. The study was approved by a local ethic committee and followed principles of the Declaration of Helsinki.

Single-blinded controlled clinical trial. The study involved stroke patients with hemiparesis (no more than 3 points on a scale Rankin). Experimental groups are determined by the target training parameter (time and general gait parameters, EMG and kinematics of leg's joints). One target parameter is using for one group. The number of sessions is 8-11 for each patient during three weeks of hospital stay. The duration of each session for each patient on each training day varies according to his well-being and current exercise tolerance, but does not exceed 30 minutes of training in one session. . Changes in biomechanical parameters that occurred at the end of the training course are assessed in comparison with those before training, and both statuses (before and after training) are compared with similar gait parameters in a group of healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Age - < 75 years;
* type of stroke - ischemic;
* structure of the lesion - cerebral hemisphere;
* disease type - primary;
* functional ability to walk for at least 5 minutes without using external means of support;
* absence of reduced higher mental functions,
* sensorimotor aphasia,
* muscle tone in the limbs above 2 points according to Ashworth (Modified Ashworth Scale);
* no history of orthopedic and neurological pathology; absence of pronounced pain syndrome

Exclusion Criteria:

* Signs of orthostatic hypotension during training,
* patient desire to withdraw from the study,
* neurological deficit worsening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Gait cycle | Change from baseline at 3 weeks
  gait cycle duration - at seconds;
Foot clearance | Change from baseline at 3 weeks
  foot clearance at centimeters;
Speed of walking | Change from baseline at 3 weeks
  walking speed - km/h;
Stance phase | Change from baseline at 3 weeks
  stance phase at percent of gait cycle duration,
Single support phase | Change from baseline at 3 weeks
  single support phase at percent of gait cycle duration
Hip joint amplitude | Change from baseline at 3 weeks
  hip joint range of motion at degree
Knee joint amplitude | Change from baseline at 3 weeks
  knee joint range of motion at degree
Ankle joint amplitude | Change from baseline at 3 weeks
  ankle joint range of motion at degree
EMG amplitude of tibialis anterior muscle | Change from baseline at 3 weeks
  envelope EMG amplitude of the tibialis anterior muscle at mkV
EMG amplitude of gastrocnemus muscle | Change from baseline at 3 weeks
  envelope EMG amplitude of the gastrocnemus muscle at mkV
EMG amplitude of quadriceps femoris muscle | Change from baseline at 3 weeks
  envelope EMG amplitude of the quadriceps femoris muscle at mkV
EMG amplitude of Hamstring muscle | Change from baseline at 3 weeks
  envelope EMG amplitude of the hamstring muscle at mkV

SECONDARY OUTCOMES:
Muscle strength | Change from baseline at 3 weeks
  Muscle strength was assessed using the MRC (Medical Research Council Weakness Scale). MRC is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction). Paresis is defined as light at compliance with strength 4 points, moderate - 3 points, pronounced - 2 points, rough - 1 point and with - 0 points.
Activities of Daily Living | Change from baseline at 3 weeks
  The Barthel Index for Activities of Daily Living where 0 is no activity and score 100 is normal activity.
Modified Rankin Scale for Neurologic Disability | Change from baseline at 3 weeks
  Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability and ranged from 0 (no symptoms) to +6 - dead.
The Timed Up and Go Test | Change from baseline at 3 weeks
  Mobility is assessed based on time to complete the test: where < 10 seconds = normal, < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid.
The Medical Research Council Weakness Scale | Change from baseline at 3 weeks
  The Medical Research Council Weakness Scale where grades: 0 is paralysis;5 - is normal.

CONTACTS AND LOCATIONS:
Overall Officials: Galina E Ivanova, PhD, Study Chair — Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency
Locations (1):
- FCCerebroPathStroke, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No